CLINICAL TRIAL: NCT05491161
Title: The Motility Mother-Child Cohort - Gut Microbes, Diet and Bowel Habits in Early Life
Brief Title: The Motility Mother-Child Cohort
Acronym: MOTILITY
Status: Active, not recruiting | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: University College Cork (Other); Technical University of Munich (Other); Quadram Institute Bioscience (Other); University of Aarhus (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Henrik Munch Roager, Associate Professor, University of Copenhagen
Other Study IDs: M241
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Diet, Healthy; Infant Development
Keywords: Microbiome; Metabolomics; Nutrition; Bowel habits
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Longitudinal study — Longitudinal study following infant development from birth to 1 year of age

SUMMARY:
The overall aim of the project is to investigate how bowel habits and nutrition in early life relate to the infant gut microbiome and metabolome from birth to 1 year of age. By unravelling links between these factors in early life, we might be able to identify new putative mechanisms by which diet via microbiota-dependent pathways affects intestinal motility in early life. Furtermore, it will be explored how the development of the gut microbiome associates with the child´s development.

DETAILED DESCRIPTION:
A cohort including 125 mother/infant pairs will be established with the purpose of following the infants' progression in diet, bowel habits, gut and oral microbiome, gut and oral metabolome, physiological and mental development from birth to 12 months of age. This will be possible by longitudinal collection and analysis of biological samples and data from birth until 1 year of age.

The primary hypotheses to be tested are that early dietary patterns (composition, complexity, quality, and timing) and bowel habits (stool frequency, consistency, and transit time) are associated with the development of the infant gut microbial composition and metabolism.

The secondary hypotheses to be tested are that the development of the infant gut microbial composition and metabolism associate with growth (body weight, length, body mass index, head circumference, body composition), development of the immune system as reflected in the gut (fecal cytokines, immunoglobulins, lipopolysaccharide, antigens) as well as the systemic circulation (blood cytokines, immune cells), host metabolism (blood metabolome, appetite hormones, urine metabolome), and physical development (sleep, motor development, mental development).

The tertiary hypotheses to be tested are that the establishment and development of the infant gut microbiome is associated with external environmental factors (household, siblings, maternal diet, maternal fecal microbiome, maternal physical activity, birth conditions, and perinatal factors), and internal factors (infant oral cavity, tooth development, use of pacifier).

ELIGIBILITY:
Mothers Inclusion Criteria:

* Age: 18-40 years of age at inclusion
* Speaking Danish (since all written and oral information will be in Danish)
* Willing to store their child's biological samples in a small closed container in their own freezer at home

Mothers Exclusion Criteria:

* Gestational age more than 34 weeks at time of recruitment
* Diagnosed with gestational diabetes during this current pregnancy
* Diagnosed with preeclampsia during this current pregnancy
* Diagnosed with any severe or chronic diseases*
* Expecting triplets or higher order of multiple pregnancy
* Concurrent participation in another study
* Not capable of following the examinations according to the investigator´s instructions

Infants Inclusion Criteria:

- Gestational age at birth: 36 weeks or later

Infants Exclusion Criteria:

- Severe chronic illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy population
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Infant gut microbiome composition | Faecal samples collected bi-weekly from birth until 12 months
  Changes in gut microbiome measured by DNA/RNA sequencing of longitudinal faecal samples from infants

SECONDARY OUTCOMES:
Infant gut metabolome | Faecal samples collected bi-weekly from birth until 12 months
  Faecal metabolome as assessed by untargeted metabolomics
Infant bowel habits | Bi-weekly from birth until 12 months
  Changes in bowel habits as measured by stool frequency, stool consistency and stool colour from birth through to 12 months of age
Infant intestinal transit time | 9 and 12 months
  Intestinal transit time estimated by sweet-corn transit time through the gastrointestinal tract
Infant dietary patterns | Bi-weekly from birth until 12 months
  Changes in dietary patterns recorded using food frequency questionnaires
Infant nutrient intake | 6, 9 and 12 months
  Assessment of dietary intake by 3-days 24-hour recall
Total faecal bacteria | Faecal samples collected bi-weekly from birth until 12 months
  Changes in total faecal bacteria as measured by quantitative PCR and flow cytometry
Infant body weight | 0, 1, 3, 6, 9, and 12 months
  Changes in body weight from birth measured in gram (g) or kilogram (kg)
Infant body length | 0, 1, 3, 6, 9, and 12 months
  Changes in body length measured in centimeters (cm)
Infant growth | 0, 1, 3, 6, 9, and 12 months
  Infant weight and length will be aggregated to determine infant growth status
Infant head circumference | 0, 1, 3, 6, 9, and 12 months
  Changes in head circumference measured in centimeters (cm)
Infant fat stores | 3, 6, 9, and 12 months
  Changes in skin folds (triceps & subscapularis) measured with a skinfold caliper
Infant body composition | 9 and 12 months
  Changes in body composition as measured by bioimpedance
Infant urine metabolome | 2 days, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 months
  Changes in urine metabolome as assessed by untargeted metabolomics

OTHER OUTCOMES:
Infant faecal short-chain fatty acids | Faecal samples collected bi-weekly from birth until 12 months
  Changes in short-chain fatty acid production as measured by targeted metabolomics
Infant blood metabolome | 3, 6, 9, and 12 months
  Changes in blood metabolome as assessed by untargeted metabolomics
Maternal breast milk metabolome | 1, 2, 3, 4, 5, and 6 months postpartum
  Changes in breast milk metabolome as assessed by untargeted metabolomics
Maternal breast milk human milk oligosaccharides | 1, 2, 3, 4, 5, and 6 months postpartum
  Changes in breast milk human milk oligosaccharides (HMOs) measured by metabolomics
Infant blood appetite hormones | 3, 6, 9, and 12 months
  Concentrations of appetite hormones in blood
Infant faecal proteome | Faecal samples collected bi-weekly from birth until 12 months
  Changes in food- and microbiota-related antigens
Infant faecal pH | Faecal samples collected bi-weekly from birth until 12 months
  Changes in faecal pH
Infant faecal oligosaccharide residues | Faecal samples collected bi-weekly from birth until 12 months
  Changes in faecal oligosaccharide residues
Infant faecal cytokines | Faecal samples collected bi-weekly from birth until 12 months
  Changes in faecal cytokines
Infant faecal immunoglobulins | Faecal samples collected bi-weekly from birth until 12 months
  Changes in faecal immunoglobulins
Infant faecal lipopolysaccharides | Faecal samples collected bi-weekly from birth until 12 months
  Changes in faecal lipopolysaccharides (LPS)
Infant blood immune cell profiles | 3, 6, 9, and 12 months
  Blood immune cell profiling
Infant blood cytokine profiles | 3, 6, 9, and 12 months
  Blood cytokine profiling
Infant gastrointestinal symptoms | Occurrence from birth until 12 months
  Gastrointestinal symptoms and related symptoms (fever, bloating, vomiting, diarrhea, constipation, irritability (crying time)) from birth through to 12 months of age
Infant general health status | 3, 6, 9, and 12 months
  General health status of the infant in relation to occurrence of any illness and health care visits for sickness, use of antibiotics and medication.
Maternal nutrient intake | Gestational week 35-37, 3 months and 9 months postpartum
  Assessment of dietary intake by 3-days 24-hours recall
Infant oral microbiome | 3, 6, 9, and 12 months
  Changes in saliva microbiome measured by DNA/RNA sequencing of saliva samples from infants
Infant oral metabolome | 3, 6, 9, and 12 months
  Changes in saliva metabolome measured by untargeted metabolomics
Infant tooth development | 3, 6, 9, and 12 months
  Infant tooth development during the first year of life
Infant sleep patterns | 3, 6, 9, and 12 months
  Infant sleep patterns during the first year of life based on the Brief Infant Sleep Questionnaire (BISQ)
Infant motor development | 3, 6, 9, and 12 months
  Infant motor development as assessed by World Health Organization (WHO) assessment of motor milestones
Mental well-being of infants | 9 and 12 months
  Infant mental health as assessed by the Copenhagen Infant Mental Health Screening (CIMHS) at 9 and 12 months of age

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Nutrition, Exercise and Sports, Copenhagen, Denmark

REFERENCES:
- [Derived] Stolberg-Mathieu G, Mikkelsen LS, Gottlieb AD, Molgaard C, Roager HM. The MOTILITY Mother-Child Cohort: a Danish prospective longitudinal cohort study of the infant gut microbiome, nutrition and bowel habits - a study protocol. BMJ Open. 2025 Jun 18;15(6):e094965. doi: 10.1136/bmjopen-2024-094965. PMID 40533209